CLINICAL TRIAL: NCT05365100
Title: A Multicenter Phase 1/2 Clinical Study to Evaluate the Safety and Efficacy of BN102 in Patients With Previously Treated Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL/SLL) and B-cell Non-Hodgkin's Lymphoma (NHL)
Brief Title: A Study of BN102 in Patients With Previously Treated CLL/SLL and B-cell NHL
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to company decision
Sponsor: BioNova Pharmaceuticals (Shanghai) LTD. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BN102-101
Record Dates: First submitted 2022-04-26; First posted 2022-05-09 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: CLL/SLL; NHL
Keywords: relapsed/refractory or intolerable
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Phase1dose escalation (Experimental): Phase1 Dose Escalation Multiple dose levels of BN102 to be evaluated; determination of MTD/Phase 2 recommended dose(RP2D)
  Interventions: Drug: BN102
- Phase2 expansion in R/R MCL with BTK inhibitor treatment history (Experimental): patients must have received at least one systemic treatment and failed or relapsed, patients previous treatment should with BTK inhibitor, approximate 12-23 patients this group
  Interventions: Drug: BN102
- Phase2 expansion in R/R MCL without BTK inhibitor treatment history (Experimental): patients must have received at least one systemic treatment and failed or relapsed, patients previous treatment should without BTK inhibitor, approximate 12-23 patients this group
  Interventions: Drug: BN102
- Phase2 expansion in R/R CLL/SLL with BTK inhibitor treatment history (Experimental): patients must have received at least one systemic treatment and failed or relapsed, patients previous treatment should with BTK inhibitor, approximate 12-23 patients this group
  Interventions: Drug: BN102
- Phase2 Expansion in R/R CLL/SLL without BTK inhibitor treatment history (Experimental): patients must have received at least one systemic treatment and failed or relapsed, patents previous treatment should without BTK inhibitor, approximate 12-23 patients this group
  Interventions: Drug: BN102
- Phase2 Expansion in other R/R B-NHL with BTK inhibitor treatment history (Experimental): patients must have received at least one systemic treatment and failed or relapsed, patents previous treatment should with BTK inhibitor, approximate 12-23 patients this group
  Interventions: Drug: BN102
- Phase2 Expansion in other R/R B-NHL without BTK inhibitor treatment history (Experimental): patients must have received at least one systemic treatment and failed or relapsed, patents previous treatment should without BTK inhibitor, approximate 12-23 patients this group
  Interventions: Drug: BN102

INTERVENTIONS:
Drug: BN102 — oral tablets: BN102, BID
  Other Names: AS-1763

SUMMARY:
This is a Multicenter Phase 1/2 Clinical Study to Evaluate the Safety and Efficacy of BN102 in Patients with Previously Treated Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL/SLL) and B-cell Non-Hodgkin's Lymphoma (NHL)

DETAILED DESCRIPTION:
The study is divided into 2 phases. Phase1 dose escalation part will enroll 17-36 patients to evaluate safety and tolerance of BN102 in patients with relapsed/refractory (R/R) CLL/SLL and B-NHL to determine maximum tolerated dose and recommended phase2 dose(RP2D).

Phase 2 expansion part will enroll 72-138 patients and be conducted at the selected dose level to further evaluate the safety and tolerability of BN102,as well as preliminary efficacy in specific subtypes of lymphoma. Patients will be allocated into 6 lymphoma subgroup cohorts depends on whether their previous treatment with or without BTK inhibitors.

* Cohort 1: patients with mantle cell lymphoma (MCL) previously treated with BTK inhibitors
* Cohort 2: patients with MCL who have not previously received a BTK inhibitor
* Cohort 3: patients with CLL/SLL who have received prior BTK inhibitors
* Cohort 4: patients with CLL/SLL who have not received prior BTK inhibitors
* Cohort 5: other B-NHL patients who have received prior BTK inhibitors
* Cohort 6: other B-NHL patients who have not received prior BTK inhibitors

Patients will receive orally administrated BN102 twice daily under fasting status. Study drug will be administered in 28-day cycles until disease progression or unacceptable toxicity, death, ICF withdraw ect. Subjects may receive study drug in the inpatient or outpatient setting.

ELIGIBILITY:
Inclusion Criteria:

All of the following conditions must be met for subject enrollment:

* Have fully understood and voluntarily signed the informed consent form ;
* Age ≥ 18 years;
* In phase 1, subjects with histologically confirmed CLL/SLL or B-cell NHL who are relapsed/refractory or intolerable after at least 1 prior line of adequate therapy, and have no better treatment choice as assessed by the investigator;
* In Phase 2, the 6 cohorts had the following specific enrollment criteria and required further treatment:
* Cohort 1: histologically confirmed MCL, failure or intolerance to at least one prior treatment including BTK inhibitor;
* Cohort 2: histologically confirmed MCL, failure or intolerance to at least 1 prior standard of care (BTK inhibitors naive);
* Cohort 3: histologically confirmed CLL/SLL, failure or intolerance to at least 1 prior treatment including BTK inhibitor;
* Cohort 4: histologically confirmed CLL/SLL, failure or intolerance to at least 1 prior standard of care (BTK inhibitors naive);
* Cohort 5: histologically confirmed other B-NHL, failure or intolerance to at least 1 prior treatment including BTK inhibitor;
* Cohort 6: histologically confirmed other B-NHL, failure or intolerance to at least 1 prior standard of care (BTK inhibitors naive);
* In addition to CLL and WM, subjects must have at least one radiographically measurable lesion
* ECOG score 0-2;
* Male or female patients of childbearing potential must agree to use effective methods of contraception

Exclusion Criteria:

* Primary central nervous system lymphoma or lymphoma involving the central nervous system;
* Serological status reflects active viral hepatitis B (HBV) or viral hepatitis C (HCV) infection
* HIV infection;
* Abnormalities in hematology lab results
* Cardiac, hepatic, renal, and coagulation abnormalities
* Concomitant clinically significant systemic active infection uncontrollable after appropriate antibiotics or other treatment;
* Expected survival of no more than 24 weeks as judged by the investigator;
* Major surgery within 4 weeks prior to the first dose of study drug
* Required or received anticoagulant therapy (warfarin, or equivalent vitamin K antagonist, or direct thrombin inhibitor, or factor Xa inhibitor, etc.) within 7 days prior to the first dose of study treatment;
* Had undergone cell transplantation or chimeric antigen receptor T cell (CAR-T) therapy within 60 days prior to enrollment
* Combined with uncontrolled active immune cytopenia
* Previous treatment with non-covalently binding BTK inhibitors (e.g. LOXO-305, MK-1026, etc.);
* Pregnant (positive pregnancy test at screening) or lactating female patients;
* QTcF > 450 msec in male patients or QTcF > 470 msec in female patients or other significant ECG abnormalities as judged by the investigator;
* Toxicities due to prior antilymphoma therapy have not stabilized and have not recovered to ≤ Grade 1 (except for clinically insignificant toxicities such as alopecia, etc.);
* History of other malignancies within 5 years prior to enrollment, special cases must be discussed with the medical monitor;
* Prior systemic anti-tumor therapy or investigational therapy received less than 4 weeks or 5 half-lives (whichever is shorter) from the start of the planned study treatment;
* Use of strong CYP3A inhibitors or inducers and proton pump inhibitors within 1 week or 5 half-lives (whichever is shorter) before administration of the first study drug;
* History of acute myocardial infarction, unstable angina, stroke, intracranial hemorrhage or transient ischemic attack within 6 months prior to enrollment; New York Heart Association (NYHA) grade 3 and 4 congestive heart failure;
* Live viral vaccination within 28 days prior to the first dose of study drug;
* Unable to take oral drugs, or have severe gastrointestinal diseases that investigator believes that it may affect the absorption of the study drug;
* Insufficient compliance of patients participating in this clinical study as judged by the investigator;
* Any other disease or condition in the judgment of the investigator that the patient is not suitable for the study drug, or will affect the interpretation of the study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07 (Estimated); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events and Clinical Laboratory Abnormalities | 2 year
  Phase1
To assess the preliminary anti-tumor activity of BN102 based on Overall response rate(ORR) assessed by the Investigator | 3 years
  Phase2

SECONDARY OUTCOMES:
Overall response rate(ORR) as assessed by the Investigator | 3 years
  Phase1
Time to response(TTR) as assessed by the Investigator | 3 years
  Phase1/2
Duration of response(DoR) as assessed by the Investigator | 3 years
  Phase1/2
Progression-free survival(PFS) as assessed by the Investigator | 3 years
  Phase1/2
Overall Survival(OS) as assessed by the Investigator | 3 years
  Phase1/2
To characterized Maximum Plasma Concentration [Cmax] of BN102 by collecting and evaluating the serum at the protocol specified time points. | at the end of cycle1(each cycle is28days) and Cycle2 Day1
  Phase1/2
To characterized Peak time(Tmax) of BN102 by collecting and evaluating the serum at the protocol specified time points. | at the end of cycle1(each cycle is28days) and Cycle2 Day1
  Phase1/2
To characterized Clearance half-life (T1/2) of BN102 by collecting and evaluating the serum at the protocol specified time points. | at the end of cycle1(each cycle is28days) and Cycle2 Day1
  Phase1/2
To characterized Area under the blood concentration-time curve (AUC0-t) of BN102 by collecting and evaluating the serum at the protocol specified time points. | at the end of cycle1(each cycle is28days) and Cycle2 Day1
  Phase1/2
To characterized Clearance rate (CL/F) of BN102 by collecting and evaluating the serum at the protocol specified time points. | at the end of cycle1(each cycle is28days) and Cycle2 Day1
  Phase1/2
To characterized apparent volume of distribution (Vd/F) of BN102 by collecting and evaluating the serum at the protocol specified time points. | at the end of cycle1(each cycle is28days) and Cycle2 Day1
  Phase1/2
To characterized mean residence time (MRT) of BN102 by collecting and evaluating the serum at the protocol specified time points. | at the end of cycle1(each cycle is28days) and Cycle2 Day1
  Phase1/2
Number of Participants with Adverse Events and Clinical Laboratory Abnormalities | 2 years
  Phase2

CONTACTS AND LOCATIONS:
Overall Officials: Weili Zhao, Prof., Principal Investigator — Shanghai Jiaotong University school of Medicine, Ruijin Hospital
Locations (6):
- China (6):
  - ZhuJiang Hospital of Southern Medical University, Guangzhou
  - The First Affiliated School of Guangxi Medical University, Nanning
  - Shanghai Jiao Tong University School of Medicine, Ruijin Hospital, Shanghai
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - Henan Oncology Hospital, Zhengzhou

IPD SHARING:
Plan to Share IPD: No